CLINICAL TRIAL: NCT02121574
Title: A Study To Determine The Accuracy Of Zero-Flux And Ingestible Thermometers In The Perioperative Setting
Brief Title: Accuracy of Zero-flux and Ingestible Thermometers
Status: Completed | Type: Observational
Sponsor: Brighton and Sussex University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Dr C. Mark Harper, Dr C. Mark Harper Consultant Anaesthetist, Brighton and Sussex University Hospitals NHS Trust
Other Study IDs: WKR0-2013-0051
Record Dates: First submitted 2014-04-22; First posted 2014-04-23 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Surgery; Hypothermia; Anesthesia
Keywords: Surgery; thermometers; Hypothermia; anesthesia; temperature
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Zero-flux and ingestible thermometer: Ingestion of a capsule thermometer pre-operatively Attachment of a zero flux temperature electrode intraoperatively Standard oesophageal thermometer
  Interventions: Device: Zero flux and ingestible thermometers

INTERVENTIONS:
Device: Zero flux and ingestible thermometers

SUMMARY:
Background When a patient is anesthetised and undergoes an operation, their body temperature falls. Managing a body temperature properly by keeping it within normal limits has been shown to improve recovery from surgery.

A vital part of managing temperature is being able to measure it properly. There are several ways of doing so, which consist of invasive methods such as temperature probes in the oesophagus and bladder, and non invasive methods such as infrared scanners and ear canal probes. During an operation, temperature changes as small as 0.5 °C can affect outcomes but, currently, only invasive methods are reliable enough to detect this. Oesophageal probes can't be used in patients who are not anaesthetised during their operations, and it is inappropriate to insert a urinary catheter should it not be otherwise needed.

The purpose of this study is to look at two new methods of measuring a patient's temperature which would help us in these situations. The first is called zero-flux thermometry and involves placing an adhesive pad to the forehead, which gives constant measurement of a patient's core temperature. The second involves swallowing an ingestible capsule that is no bigger than a normal pill. This technique has been very useful in research tracking a patient's core temperature as they are transferred through different areas over a longer period of time. Whilst these two methods are potentially very useful, they have never been tested on hospital patients.

Aims:

The investigators want to determine whether readings from these thermometers are accurate enough to be used in patients before, during and after surgery. Should they prove to be sufficiently accurate it will allow us to improve patient care through both clinical practice and research.

Plan:

During operations, temperature is routinely measured in line with NICE guidelines with a thermometer placed in the nose or oesophagous. The investigators will not be changing routine practice in any way, but checking measurements from the new devices against the proven, routine ones.

The investigators plan to record measurements from each device every minute throughout the operation in 20 patients. The investigators will then perform statistical tests to check their accuracy.

Study Hypothesis: Zero flux and ingestible thermometers are not significantly different at detecting patients body temperature than oesophageal temperature probes

DETAILED DESCRIPTION:
Summary:

The study has been designed to provide information on the suitability and accuracy of two methods of temperature measurement in the perioperative period.

Background:

Good perioperative temperature management is an important means of improving patient outcome [1].

An essential part of optimal management is accurate temperature measurement. The gold standard is pulmonary artery catheter (PAC) measurement. However, these are used infrequently in British practice due to the high rates of associated complications. Urinary bladder and oesophageal temperatures are sufficiently accurate but are unsuitable for many patients [2]. For example it is not possible to use oesophageal probes in awake patients and many patients are not catheterised.

Although non-invasive and relatively cheap means of measuring temperature (such as aural canal probes and infrared scanners) exist, they are neither accurate nor consistent enough to distinguish the 0.5˚C differences which have a significant effect on patient outcomes [2].

In this study, the investigators plan to look at two methods of temperature measurement which potentially offer significant improvements to surgical care.

The first is a new method known as zero-flux thermometry. This is completely non-invasive, involving no more than placing an adhesive pad to the forehead. Connected up to a monitor, this will equilibrate with the patient's core temperature and give a constant read-out.

The second is an ingestible capsule. These have become an important tool for measuring both hypothermia and hyperthermia in other settings. Their accuracy has not, however, been tested in hospital patients. This technology, although too expensive for routine use, offers significant advantages for research as they can provide a constant record of temperature throughout the patient's stay in hospital. For example, the investigators' audit data show that if patients admitted with fractured neck of femur become hypothermic at any time, their mortality increases. Subsequent to this we showed that patient temperatures drop significantly between ambulance, A&E and admission to the ward. These parts of the patient journey are possible targets for the prevention of hypothermia and the continuous monitoring offered by these devices will allow us to accurately test the efficacy of the interventions.

Aims and objectives:

The aim of this study is to determine the accuracy in the perioperative period of zero-flux and ingestible temperature readings.

Previous studies have shown that oesophageal and nasopharyngeal measurements can be taken as an accurate reflection of core temperature [2]. The consistency and accuracy of the other two will be compared to this.

Plan of investigation:

This study will be purely observational. There will be no interference with current practice. Nasopharyngeal/oesophageal probes are routinely placed, according to NICE guidelines, in these patients. The zero-flux thermometer is non-invasive and the ingestible capsule no bigger than a pill, so neither provide any additional risk to the patient.

Temperature readings will be downloaded from each of the three devices with a maximum interval of 1 minute. The investigators have calculated that readings from 15 subjects will provide sufficient power. The investigators plan to recruit 20 patients. Analysis of agreement between the methods will be performed as suggested by Bland and Altman[3].

ELIGIBILITY:
Inclusion Criteria:

Participants will be patients undergoing elective gynaecological, vascular or urological surgery at the Royal Sussex County Hospital, and as such will be seen at a pre-operative assessment clinic as part of their normal work up for theatre.

Exclusion Criteria:

* Lacking mental capacity
* Not speaking English
* Malignancy in medical history
* Undergoing open abdominal surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be patients undergoing elective gynaecological, vascular or urological surgery at the Royal Sussex County Hospital, and as such will be seen at a pre-operative assesment clinic as part of their normal work up for theatre.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Comparing the accuracy of zero flux and ingestible thermometers to oesophageal temperature probes. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: James M Jack, MBBS BSc, Principal Investigator — BSUH NHS Trust
Locations (1):
- Royal Sussex County Hospital, Brighton, East Sussex, United Kingdom

REFERENCES:
- [Derived] Jack JM, Ellicott H, Jones CI, Bremner SA, Densham I, Harper CM. Determining the accuracy of zero-flux and ingestible thermometers in the peri-operative setting. J Clin Monit Comput. 2019 Dec;33(6):1113-1118. doi: 10.1007/s10877-019-00252-9. Epub 2019 Jan 8. PMID 30623279